CLINICAL TRIAL: NCT04774588
Title: Holographic Streaming of Input From Video Capture Devices During Interventional Radiology Procedures - a Feasibility Study (Hololens Study)
Brief Title: HoloStream Study - Video Capture Device Usage
Acronym: Holo-Stream
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Darshan Bakshi, Interventional Radiologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB21-0111
Record Dates: First submitted 2021-02-08; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Nephrostomy; Complications; Fistula; Central Venous Catheter Thrombosis
MeSH Terms: conditions — Fistula; Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Intervention Model Description: Methodology:
  Single center randomized controlled pilot feasibility study. Firstly, VSI streamer software will be used for real time streaming of input from the fluoroscopy unit to a Head mounted display (Hololens 2) worn by the operator. This will be utilized to perform angiographic procedures on a 3D vascular model. Mock benchtop
  angiographic catheterization procedures will be performed in order to ensure practicality, safety and initial usability.
  Subsequently, appropriate patients undergoing elective Interventional Radiology procedures will be screened and enrolled. After performing these procedures on the first two patients, procedural parameters will be reviewed and subsequent patients will be enrolled if no safety concerns have arisen in the first two patients. Patients will be enrolled until a total of 60 procedures have been performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using VSI Streamer and Telemedicine Study (Other): Using the real time streaming of input from video capture devices to a head mounted display during interventional radiology procedures
  Interventions: Other: VSI streamer and Microsoft Hololens 2 classed as a Class III device by Health Canada.
- Not using VSI Streamer and Telemedicine Study (Placebo Comparator): Not using real time streaming of input from video capture devices to a head mounted display and just using current standard imaging in the Interventional Suite.
  Interventions: Other: VSI streamer and Microsoft Hololens 2 classed as a Class III device by Health Canada.

INTERVENTIONS:
Other: VSI streamer and Microsoft Hololens 2 classed as a Class III device by Health Canada. — 1.1 Description of VSI streamer device and software The VSI Streamer is a box that can be connected to ultrasound, endoscope, microscope, laparoscope and other devices via HDMI connection. The view of the imaging devices, which is conventionally displayed on a monitor, is transmitted wirelessly and in real time to the Mixed Reality HoloLens 2 (Microsoft Inc.) and appears as a virtual monitor that can be flexibly moved and positioned in space. Since this is Mixed Reality, the real environment remains visible. If required, several virtual monitors can be streamed into the Mixed Reality glasses at the same time

SUMMARY:
Objectives:

Primary

* Evaluate the primary operator usability of VSI streaming software for realtime streaming of images from video capture devices to a head mounted display (Hololens 2) during Interventional Radiology procedures Secondary
* Evaluate Radiographer usability of VSI streaming software.
* Develop suggestions for future research studies to assess the safety and efficacy of the VSI streamer software during other Interventional radiology procedures
* Evaluate the impact of VSI streaming software on room setup time, procedural time and fluoroscopy time
* Assess the feasability of remote collaboration by real time image transmission between remote devices through 3D telemedicine

DETAILED DESCRIPTION:
The ergonomic design and setup of an operating/procedure room have long been a studied topic of interest. Back in 1999, an article (1) reviewed the ongoing research into the effects that operator posture, the operating room environment, and visualization of screens have on the ergonomics of surgery. They made the observation that 'future efforts to create a more user- friendly operating room environment will require the rethinking of traditional concepts of architecture, asepsis, and staffing (1). As technology rapidly advances, we are increasingly able to reassess and enhance the current ergonomic structure and setup of operating rooms and procedures.

Interventional radiology (IR) refers to a variety of minimally invasive procedures using small- caliber catheters under fluoroscopic or ultrasound guidance for the treatment of vascular and urologic, gastrointestinal conditions without the need for open surgery (2).

Interventional Radiology has the unique ergonomic consideration of the placement of the intraoperative viewing monitors (3). To perform any Interventional Radiology procedure, radiologists currently use a ceiling mounted or floor mounted image intensifier, a ceiling mounted screen and a small floor mounted monitor. In many procedures (usually those requiring downstream access into the vessel, arm or neck vascular access) the Radiologist has to move their own position to visualize all the screens, as it is impossible to rotate the screens adequately so that they are in a direct line with the Radiologists vision. Previous studies of office video terminal display (VDT) users demonstrate that the preferred viewing angle for VDTs is between 10° to 25° below the line of sight(4). The monitors are placed in such a way that the Interventional radiologist cannot possibly maintain the correct line of sight without some neck movement and craning. Inevitably, long periods of time standing in this awkward position can lead to musculoskeletal issues for the radiologist, as well as the stress of performing a procedure safely without the best line of vision.

The Interventional Radiologist is also wearing a heavy lead apron during the procedure, which adds to the ergonomic challenges. The incidence of neck and back pain increases with hours of apron use and years of practice, and may be the result of a combination of axial load (ie, prolonged standing in protective garments), awkward or poor posture (necessitated by leaning or bending to accomplish procedures), and repetitive injury accumulated over years of practice. (5)

In addition, there are multiple other screens monitoring patient parameters which are outside of the Interventional radiologist's field of view during the procedure, creating further safety concerns. Of note, other current concerns in the Interventional suite are costly screen breakage during manoeuvre of the screens during suite setup, and sterility issues that arise when the monitor is brought too close to the operating field.

The intention is that the new device will project a hologram of all the screens which can be positioned exactly in front of the operator at all times, irrespective of the patient position. Because it is mixed reality, the operator can still see their surroundings and perform the procedure exactly as normal.

With this technology, multiple screens of different modalities can be added, such as CT scans, MRI scans and 3D rendered holograms. Specific device instructions can also be visualized if necessary, without the requirement for the radiologist to leave the sterile procedure site.

The device can also be used to stream fluoroscopic and 3D images to a remote hololens or computer screen. This can be utilized for remote assistance and mentoring purposes. It will also be especially useful in the context of COVID-19, where reducing the clinical exposure of health care workers is of vital importance.

The main intention of the pilot study is to assess whether the hypothesis that the VSI streamer and HMD will indeed improve the ergonomics of the interventional suite sufficiently enough that the Interventional radiologist can perform the procedures more comfortably and safely. The practicalities of adding the VSI Streamer and HMD to the interventional suite setup will also be assessed.

During this initial pilot study, a practical assessment will be performed of the usability of the VSI streamer during commonly performed elective angiographic procedures. This will identify which procedures are particularly suited to this technology.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring the following elective outpatient angiographic procedure are eligible for this study.

These procedures include Nephrostomy tube replacement, Central venous access for line placement, Upper limb fistula access for angiography and associated procedures such as angioplasty or stent insertion, antegrade or retrograde Common Femoral Arterial access for angiography and associated procedures such as angioplasty or stent insertion.

All patients must be 18 years of age or older.

All patients must be able to provide written informed consent

Exclusion Criteria:

* Patients unable to provide written consent. Patients unwilling to provide written consent.

Research participation is not in the best interest of the patient.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the usability and effectiveness of VSI streaming software | 1 year
  • Evaluate the operator usability of VSI streaming software for realtime streaming of images from video capture devices to a head mounted display (Hololens 2) during Interventional Radiology procedures The NASA TLX questionnaire will be used to assess operator usability and effectiveness. Total score of the questionnaire items will be reported as medians and interquartile ranges and compared using non parametric Kruskal-Wallis and Mann-Whitney U tests as appropriate.

IPD SHARING:
Plan to Share IPD: No